CLINICAL TRIAL: NCT03176277
Title: A Phase I/II Open Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Clinical Efficacy of ONO-7475 in Patients With Acute Leukemias or Myelodysplastic Syndromes
Brief Title: A Study of ONO-7475 in Patients With Acute Leukemias
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Protocol defined futility criteria
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7475-01
Record Dates: First submitted 2017-05-19; First posted 2017-06-05 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Acute Leukemia; Myelodysplastic Syndromes
Keywords: Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; MER; MERTK; TYRO3; AXL; AML; Relapsed/ Refractory AML; TAM; MDS; Myelodysplastic Syndrome; Relapsed/ Refractory MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: Part A: ONO-7475 open-label, dose escalation in R/R AML or R/R MDS Part D: ONO-7475 plus venetoclax open-label, dose escalation in R/R AML
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ONO-7475 3mg once daily (Experimental): Part A Initial dose level
  Interventions: Drug: ONO-7475 3mg once daily
- ONO-7475 6mg once daily (Experimental): Part A 2nd dose level
  Interventions: Drug: ONO-7475 6mg once daily
- ONO-7475 10mg once daily (Experimental): Part A 3rd dose level
  Interventions: Drug: ONO-7475 10mg once daily
- ONO-7475 6mg + Venetoclax (70-400mg) (Experimental): Part D ONO-7475 + Venetoclax combination
  Interventions: Drug: ONO-7475 6mg + Venetoclax (70-400mg)

INTERVENTIONS:
Drug: ONO-7475 3mg once daily — Part A initial dose level
  Other Names: Part A initial dose level
  Arms: ONO-7475 3mg once daily
Drug: ONO-7475 6mg once daily — Part A 2nd dose level
  Other Names: Part A 2nd dose level
  Arms: ONO-7475 6mg once daily
Drug: ONO-7475 10mg once daily — Part A 3rd dose level
  Other Names: Part A 3rd dose level
  Arms: ONO-7475 10mg once daily
Drug: ONO-7475 6mg + Venetoclax (70-400mg) — Part D ONO-7475 + Venetoclax Combination
  Other Names: ONO-7475 + Venetoclax Combination
  Arms: ONO-7475 6mg + Venetoclax (70-400mg)

SUMMARY:
[Updated]: To assess the safety and tolerability of ONO-7475 monotherapy in patients with relapsed or refractory acute myeloid leukemia or relapsed or refractory myelodysplastic syndromes and to assess: i) safety and tolerability and ii) preliminary efficacy of the combination of ONO-7475 and venetoclax in patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
Part A is a dose escalation study of ONO-7475 in patients with acute myeloid leukemia or relapsed or refractory myelodysplastic syndromes.

Part D is a dose escalation study of ONO-7475 in combination with venetoclax. ONO-7475 starting dose is selected following safety and tolerability outcome of Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years at time of screening.
2. Written informed consent by the patient (or their legal representative) prior to admission to this study. In addition, any locally required authorization (Health Insurance Portability and Accountability Act in the US), must be obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
3. Adequate renal and hepatic function defined as:

   1. Total bilirubin within 1.5 x upper limit of normal (ULN), except those with Gilberts syndrome for whom this must be ≤3 x ULN
   2. AST and ALT ≤2.5 x ULN
   3. Calculated creatinine clearance ≥45 mL/min
   4. Serum albumin ≥2.5 g/dL For any patient with laboratory values outside the ranges outlined above that are considered due to the patient's underlying disease (AML or MDS), the patient may be enrolled into the study following consultation between the Investigator and the Sponsor's Medical Officer, if the patient is likely to benefit from receiving ONO-7475 (based on the Investigator's assessment).
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 as assessed during the screening period and then again anytime during the 2-day period immediately preceding the start of dosing in Parts A and D.
5. Life expectancy of at least 3 months
6. Sexually active female patients of childbearing potential and sexually active male patients must agree to use an effective method of birth control (e.g., barrier methods with spermicides, oral or parenteral contraceptives and/or intrauterine devices) during the entire duration of the study and for 4 months after final administration of study drug. Note that sterility in female patients must be confirmed in the patients' medical records and be defined as any of the following: surgical hysterectomy with bilateral oophorectomy, bilateral tubular ligation, natural menopause with last menses >1 year ago, radiation-induced oophorectomy with last menses >1 year ago, chemotherapy-induced menopause with last menses >1 year ago.
7. Diagnosis of AML or MDS according to WHO criteria 2016 (Part A only).
8. Either criterion is met (Part A only):

   1. Patients with R/R AML with at least 5% blasts by BM biopsy or aspirate, or at least 1% blasts in peripheral blood, not likely to benefit from standard salvage chemotherapy
   2. Patients with R/R MDS who are either not eligible for (or unlikely to benefit from) other forms of therapy, including HSCT, according to the treating Physician/Investigator .
9. All patients must have received at least one previous line of therapy (Part A only).
10. Diagnosis of AML according to WHO criteria (2016) (Part D only).
11. Patients with R/R AML who have no standard-of-care options known to provide clinical benefit in patients with R/R AML (Part D only)

    1. Refractory AML: Patients who have not achieved complete remission after two cycles of induction chemotherapy (i.e., anthracycline containing regimen), four cycles of hypomethylating agents, or two cycles of other AML therapy
    2. Relapsed AML: Patients who have ≥5% BM blasts in BM, or reappearance of blasts in the peripheral blood not attributable to another cause (e.g., recovery of normal cells following chemotherapy-induced aplasia) or (re)appearance of extramedullary disease after CR of prior AML therapy.
12. Patients must have measured BM aspirate blast counts at Screening. Where the aspirate is hypo cellular or inaspirable a biopsy would be considered.
13. Patients who were refractory to or relapsed after their 1st line treatment for AML must have received 2 or less additional lines of intensive / aggressive chemotherapy, which also includes a venetoclax-based regimen, as per the latest National Comprehensive Cancer Network (NCCN) Guidelines.

Exclusion Criteria:

1. Patients with active central nervous system leukemia.
2. QT interval corrected according to Fredericia's formula (QTcF) prolongation defined as a QTcF interval >470 msec or other significant ECG abnormalities including second degree (type II) or third degree atrioventricular block or bradycardia (ventricular rate <50 beats/min).
3. Clinically significant liver disease, including active viral or other hepatitis, current alcohol abuse, or severe cirrhosis.
4. Human immunodeficiency virus (HIV), active hepatitis B (HBV) or C (HCV) infection.
5. Retinal disease (e.g., retinitis pigmentosa including Mertk mutations), retinal hemorrhage or any disorder which may inhibit follow up for retinal toxicity.
6. Serious intercurrent medical or psychiatric illness that will prevent participation or compliance with study procedures, including serious active infection (including COVID-19).
7. Acute promyelocytic leukemia (the French-American-British M3 classification).
8. Patients not recovered to Grade 1 or stabilized from the effects (excluding alopecia) of any prior therapy for their malignancies.
9. Concurrent treatment with other investigational drugs.
10. Daily requirement of ≥10 mg/day of prednisone or equivalent dose of other corticosteroids.
11. Prior HSCT within 12 weeks of the first dose of study treatment or ongoing immunosuppressive therapy for graft-versus-host disease.
12. Participation in another clinical trial with any investigational drug within 14 days or with any licensed drug within five half-lives, prior to the first ONO-7475 dosing (for Part A) or prior to the first venetoclax dosing (for Part D).
13. Prior AML or MDS therapy (non-experimental) within 14 days or 5 half-lives, whichever is longer, prior to the first dose of ONO-7475 (for Part A) or prior to the first venetoclax dosing (for Part D) (except those permitted in Section 7.1) and no residual toxicity from the prior therapy hindering of the ONO-7475 dosing (for Part A) or ONO-7475 plus venetoclax dosing (for Part D).
14. Prior radiotherapy within 21 days of screening, with the exception of localized palliative radiotherapy.
15. Patients undergoing current treatments for other cancers.
16. Pregnant or lactating women.
17. Proliferative disease (white blood cell [WBC] counts >30 x 10e9/L) confirmed prior to the first dose of ONO-7475 (for Part A) or WBC >25 x 10e9/L in Part D.
18. Active malignancy, other than AML (Parts A and D) or MDS (Part A), requiring systemic therapy except for those patients who have been diagnosed with either prostate or breast cancer and who have received a stable dose of hormone therapy for a minimum of 6 months prior to entering this study.
19. Known hypersensitivity to venetoclax (Part D only).
20. Calculated creatinine clearance <45 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (16):
- United States (16):
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, California
  - Yale University School of Medicine - Yale Cancer Center, North Haven, Connecticut
  - University of Florida (UF) - Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - The Winship Cancer Institute Emory University, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Weill Medical College of Cornell University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - The Ohio State University (OSU), Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina - Hollins Cancer Center, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kasner MT, Courtenay-Luck N, DiNardo C, Post SM, Baratam P, Magrath GN, Nakamura T, Fujii A, Prados S, Honda N, Mcbride M, Edwards-Holmes P, Stuart R. Anexelekto (Axl)/Mer Inhibitor Tamnorzatinib in Patients with Relapsed/Refractory Acute Myeloid Leukaemia: Results from a Phase I (Monotherapy) and Phase II (Combination with Venetoclax) Clinical Study. Acta Haematol. 2025 Dec 12:1-11. doi: 10.1159/000549340. Online ahead of print. PMID 41385448

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A study: a total of 29 participants signed informed consent form and were enrolled in the study. 9 participants were screen failures who did not meet eligibility criteria. 20 participants received at least 1 dose of study drug.
  Part D study: a total of 33 participants signed informed consent form and were enrolled in the study. 11 participants were screen failures who did not meet eligibility criteria. 22 participants received at least 1 dose of study drug. No dose escalation conducted.
Groups:
- ONO-7475 3mg: Part A initial dose level
- ONO-7475 6mg: Part A 2nd dose level
- ONO-7475 10mg: Part A 3rd dose level
- ONO-7475 6mg + Venetoclax: Part D combination ONO-7475 + Venetoclax
Period: Part A Dose Escalation Study
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg | ONO-7475 6mg + Venetoclax
Started | 10 | 3 | 7 | 0 (It is not applicable to Part A Dose Escalation Study.)
Completed | 0 | 0 | 0 | 0
Not Completed | 10 | 3 | 7 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 1 | 0
Not completed — Progressive disease | 3 | 1 | 3 | 0
Period: Part D ONO-7475 6mg + Venetoclax
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg | ONO-7475 6mg + Venetoclax
Started | 0 (It is not applicable to Part D combination ONO-7475 + Venetoclax study.) | 0 (It is not applicable to Part D combination ONO-7475 + Venetoclax study.) | 0 (It is not applicable to Part D combination ONO-7475 + Venetoclax study.) | 22
Completed | 0 | 0 | 0 | 22
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set, respective of Part A and Part D study.
Groups:
- ONO-7475 6mg + Venetoclax: Part D combination of ONO-7475 + Venetoclax
- Total: Total of all reporting groups
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg | ONO-7475 6mg + Venetoclax | Total
Number analyzed (Participants) | 10 | 3 | 7 | 22 | 42
Age, Continuous [Median (Full Range); unit: years]
  Age | 56.0 [23 to 77] | 65.0 [58 to 81] | 72.0 [63 to 77] | 65.5 [48 to 82] | 67.0 [23 to 82]
Age, Customized [Count of Participants; unit: Participants]
  <=60 years | 5 | 1 | 0 | 9 | 15
  >60 years | 5 | 2 | 7 | 13 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 4 | 9 | 22
  Male | 4 | 0 | 3 | 13 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 9 | 3 | 7 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 4 | 9
  White | 5 | 2 | 5 | 15 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 3 | 7 | 22 | 42
ECOG performance status [Count of Participants; unit: Participants] — Grade 0 Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Grade 2 Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  Grade 3 Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours.
  Grade 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair.
  Grade 5 Dead.
  Participants
    Grade 0 | 2 | 0 | 1 | 1 | 4
    Grade 1 | 7 | 2 | 4 | 19 | 32
    Grade 2 | 1 | 1 | 2 | 2 | 6
Height [Median (Full Range); unit: Centimeter] | 158.0 [152 to 180] | 160.0 [156 to 168] | 163.0 [155 to 173] | 168 [144 to 188] | 165 [144 to 188]
Weight [Median (Full Range); unit: Kilogram] | 76.30 [45.9 to 104.0] | 82.50 [59.1 to 102.5] | 64.10 [61.4 to 80.7] | 75.45 [39.3 to 123.6] | 74.25 [39.3 to 123.6]
BMI [Median (Full Range); unit: Kilogram per square meter] | 29.25 [19.3 to 35.2] | 32.22 [24.3 to 36.3] | 25.54 [21.2 to 27.9] | 24.03 [18.4 to 38.4] | 25.56 [18.4 to 38.4]
AML FAB classification at initial diagnosis [Count of Participants; unit: Participants] — AML FAB classification. FAB=French-American-British
  Participants
    M1 - ACUTE MYELOBLASTIC LEUKEMIA WITH MINIMAL MATURATION | 1 | 0 | 1 | 1 | 3
    M2 - ACUTE MYELOBLASTIC LEUKEMIA WITH MATURATION | 3 | 1 | 1 | 4 | 9
    M5 - ACUTE MONOCYTIC LEUKEMIA | 1 | 1 | 1 | 0 | 3
    M7 - ACUTE MEGAKARYOBLASTIC LEUKEMIA | 0 | 1 | 0 | 1 | 2
    UNKNOWN | 4 | 0 | 4 | 8 | 16
    MISSING | 1 | 0 | 0 | 0 | 1
    Acute Myeloid Leukaemia With Cup Like Morphology | 0 | 0 | 0 | 1 | 1
    M0 - Undifferentiated Acute Myeloblastic Leukemia | 0 | 0 | 0 | 5 | 5
    M4 - Acute Myelomonocytic Leukemia | 0 | 0 | 0 | 2 | 2
AML classification at initial diagnosis 2008 2016 revisions to 2008 WHO classification [Count of Participants; unit: Participants]
  ACUTE MEGAKARYOBLASTIC LEUKEMIA | 0 | 1 | 0 | 1 | 2
  ACUTE MONOBLASTIC/MONOCYTIC LEUKEMIA | 0 | 0 | 1 | 0 | 1
  ACUTE MYELOID LEUKEMIA WITH MYELODYSPLASIA-RELATED CHANGES | 3 | 0 | 1 | 9 | 13
  ACUTE MYELOMONOCYTIC LEUKEMIA | 0 | 1 | 0 | 2 | 3
  AML WITH INV(16)(P13.1Q22) OR T(16;16)(P13.1;Q22); CBFB-MYH11 | 1 | 0 | 0 | 0 | 1
  AML WITH MATURATION | 2 | 0 | 0 | 1 | 3
  AML WITH MINIMAL DIFFERENTIATION | 1 | 0 | 2 | 0 | 3
  AML WITH MUTATED RUNX1 | 0 | 0 | 1 | 2 | 3
  AML, NOS | 1 | 1 | 1 | 5 | 8
  UNKNOWN | 2 | 0 | 1 | 1 | 4
  AML Without Maturation | 0 | 0 | 0 | 1 | 1
Extramedullary involvement at diagnosis [Count of Participants; unit: Participants]
  No | 9 | 3 | 7 | 19 | 38
  Unknown | 1 | 0 | 0 | 3 | 4
AML classification performed according to WHO criteria 2016 completed at screening [Count of Participants; unit: Participants]
  ACUTE MEGAKARYOBLASTIC LEUKEMIA | 0 | 1 | 0 | 1 | 2
  ACUTE MYELOBLASTIC/MONOCYTIC LEUKEMIA | 0 | 0 | 1 | 0 | 1
  ACUTE MYELOID LEUKEMIA WITH MYELODYSPLASIA-RELATED CHANGES | 5 | 0 | 0 | 6 | 11
  ACUTE MYELOMONOCYTIC LEUKEMIA | 0 | 1 | 0 | 2 | 3
  AML WITH INV(16)(P13.1Q22) OR T(16;16)(P13.1;Q22); CBFB-MYH11 | 1 | 0 | 0 | 0 | 1
  AML WITH MATURATION | 2 | 0 | 0 | 1 | 3
  AML WITH MINIMAL DIFFERENTIATION | 1 | 0 | 3 | 0 | 4
  AML WITH MUTATED RUNX1 | 0 | 0 | 1 | 3 | 4
  AML, NOS | 1 | 1 | 2 | 7 | 11
  AML With Recurrent Genetic Abnormalities | 0 | 0 | 0 | 2 | 2
Extramedullary involvement at present [Count of Participants; unit: Participants]
  No | 9 | 0 | 0 | 22 | 31
  Unknown | 1 | 3 | 7 | 0 | 11
  Yes | 0 | 0 | 0 | 0 | 0
Current AML status [Count of Participants; unit: Participants]
  De novo | 1 | 0 | 0 | 0 | 1
  Refractory | 6 | 3 | 5 | 9 | 23
  Relapsed | 3 | 0 | 2 | 13 | 18
Immunophenotyping results available [Count of Participants; unit: Participants]
  CD34+ | 1 | 0 | 0 | 0 | 1
  Other | 8 | 3 | 7 | 17 | 35
  Missing | 1 | 0 | 0 | 5 | 6
HLA-DR results available [Count of Participants; unit: Participants] — HLA: Human Leukocyte Antigen
  Participants
    Positive | 9 | 3 | 7 | 18 | 37
    Negative | 1 | 0 | 0 | 0 | 1
    Missing | 0 | 0 | 0 | 4 | 4
HLA-DR risk group [Count of Participants; unit: Participants] — Population: This data was not captured for Part D ONO-7475 6mg + venetoclax
  Participants
    number analyzed (Participants) | 10 | 3 | 7 | 0 | 20
    Favorable | 1 | 0 | 0 | 0 | 1
    Intermediate | 2 | 0 | 1 | 0 | 3
    Adverse | 6 | 3 | 6 | 0 | 15
    Missing | 1 | 0 | 0 | 0 | 1
Left ventricular ejection fraction (LVEF) [Median (Full Range); unit: Percent] | 57.0 [41 to 74] | 62.0 [61 to 65] | 61.0 [57 to 77] | 60.0 [25 to 72] | 60.0 [25 to 77]
Time from initial diagnosis to first dose of ONO-7475 [Median (Full Range); unit: Months] | 24.3 [0.5 to 40.4] | 17.7 [11.6 to 18.4] | 12.2 [2.0 to 56.9] | 12.1 [2.0 to 81.0] | 14.7 [0.5 to 81.0]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (Part A)
Description: Incidence of most common (frequency of >20%) treatment-emergent adverse events (TEAEs) of CTCAE grade 3 or higher by preferred terms coded with MedDRA version 23.1.
  CTCAE = Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From start of study drug up to 30 days after permanent discontinuation of study drug or initiation of new anti-cancer therapy, whichever occurs first (maximum of 32 months).
Population: Safety analysis set, in participants who received at least 1 dose of ONO-7475.
Measure: Count of Participants; unit: Participants
Groups:
- ONO-7475 10 mg: Part A 3rd dose level
- Total: Part A total
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10 mg | Total
Number analyzed (Participants) | 10 | 3 | 7 | 20
Participants
  Anaemia | 4 | 1 | 2 | 7
  Febrile neutropenia | 2 | 1 | 4 | 7
  Pneumonia | 4 | 1 | 0 | 5

2. Primary Outcome: Incidence of Serious Adverse Events (Part A)
Description: Incidence (frequency ≥ 2 participants) of serious treatment-emergent adverse events (all CTCAE grades) by preferred terms coded with MedDRA version 23.1.
  CTCAE = Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: as for outcome 1
Population: Safety analysis set, in participants who received at least 1 dose of ONO-7475.
Measure: Count of Participants; unit: Participants
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg | Total
Number analyzed (Participants) | 10 | 3 | 7 | 20
Participants
  Pneumonia | 3 | 1 | 0 | 4
  Sepsis | 3 | 1 | 0 | 4
  Febrile neutropenia | 2 | 1 | 4 | 7
  Klebsiella bacteraemia | 2 | 0 | 0 | 2

3. Primary Outcome: Clinically Significant Changes in Ophthalmology Examination Parameters (Part A)
Description: Incidence (all participants) of ophthalmological treatment-emergent adverse events (all CTCAE grades) by preferred terms coded with MedDRA Version 23.1.
  CTCAE = Common Terminology Criteria for Adverse Event version 4.03.
Time Frame: as for outcome 1
Population: Safety analysis set, in participants who received at least 1 dose of ONO-7475.
Measure: Count of Participants; unit: Participants
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg | Total
Number analyzed (Participants) | 10 | 3 | 7 | 20
Participants
  Cataract cortical | 0 | 0 | 1 | 1
  Conjunctival haemorrhage | 0 | 0 | 1 | 1
  Eyelid ptosis | 1 | 0 | 0 | 1
  Night blindness | 1 | 0 | 0 | 1
  Retinal aneurysm | 0 | 1 | 0 | 1
  Retinal thickening | 1 | 0 | 0 | 1
  Retinopathy | 1 | 0 | 0 | 1
  Scleral haemorrhage | 0 | 1 | 0 | 1
  Vision blurred | 1 | 0 | 0 | 1
  Vitreous floaters | 1 | 0 | 0 | 1

4. Primary Outcome: Clinically Significant Changes in 12-Lead Electrocardiogram Parameters (Part A)
Description: Participants with clinically significant changes in 12-lead Electrocardiogram (ECG) parameters.
Time Frame: as for outcome 1
Population: Safety analysis set, in participants who received at least 1 dose of ONO-7475.
Measure: Count of Participants; unit: Participants
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg | Total
Number analyzed (Participants) | 10 | 3 | 7 | 20
Participants
  Participants with clinically significant changes in 12-lead ECG parameters | 0 | 0 | 0 | 0
  Participants without clinically significant changes in 12-lead ECG parameters | 10 | 3 | 7 | 20

5. Primary Outcome: Incidence of Adverse Events (Part D)
Description: Incidence of most common (frequency > 20%) treatment-emergent adverse events (TEAEs) of CTCAE grade 3 or higher by preferred term coded with MedDRA version 23.1.
  CTCAE = Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From start of study drug up to 30 days after permanent discontinuation of study drug or initiation of new anti-cancer therapy, whichever occurs first (maximum of 21 months).
Population: Safety analysis set, in participants who received at least 1 dose of ONO-7475 and/or venetoclax.
Measure: Count of Participants; unit: Participants
Groups:
- ONO-7475 6mg + Venetoclax: Part D ONO-7475 + venetoclax group
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 22
Participants
  Febrile neutropenia | 7
  Anaemia | 5
  Thrombocytopenia | 5

6. Primary Outcome: Incidence of Serious Adverse Events (Part D)
Description: Incidence (frequency ≥ 2 participants) of serious treatment-emergent adverse events (all CTCAE grades) by preferred terms coded with MedDRA version 23.1.
  CTCAE = Common Terminology Criteria for Adverse Events (CTXAE) Version 4.03.
Time Frame: as for outcome 5
Population: Safety analysis set, in participants who received at least 1 dose of ONO-7475 and/or venetoclax.
Measure: Count of Participants; unit: Participants
Groups:
- ONO-7475 6 mg + Venetoclax: Part D ONO-7475 6 mg + Venetoclax
Arm/Group | ONO-7475 6 mg + Venetoclax
Number analyzed (Participants) | 22
Participants
  Sepsis | 3
  Febrile neutropenia | 7
  Gastrointestinal haemorrhage | 2

7. Primary Outcome: Complete Response (CR) / Complete Response With Partial Hematologic Recovery (CRh) Rate (Part D)
Description: Summary of complete response (CR) and complete response with partial hematologic recovery (CRh) rate.
Time Frame: From baseline up to maximum of 21 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Groups:
- ONO-7475 6mg + Venetoclax: Part D ONO-7475 + venetoclax
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 22
Participants
  Complete remission | 0
  Complete response with partial hematologic recovery | 0

8. Secondary Outcome: Determination of Maximum Tolerated Dose (MTD) by Assessing Dose Limiting Toxicities (DLT) (Part A)
Description: Dose Limiting Toxicities (DLT) Criteria: 1) ONO-7475-related ≥Grade 4 hematologic toxicity, 2) any pre-existing condition that worsens by more than 1 grade or to Grade 4, not caused by AML, 3) any ≥Grade 3 non-hematologic toxicity not caused by AML (exception: alopecia, nausea, vomiting, fatigue, headache, chills, electrolyte disturbances), 4) ≥Grade 2 blurred vision (confirmed by loss of 15 letters or more on Early Treatment Diabetic Retinopathy chart and by ophthalmological and retinal assessments) not caused by AML, 5) ≥Grade 2 clinically significant changes in night blindness not caused by AML, 6) ≥Grade 3 differentiation syndrome, 7) death not caused by AML, and 8) any other event determined by the Safety Review Committee for dosing stop.
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 was applied for toxicity grading.
Time Frame: 28 days
Population: Analysis set included participants evaluable for DLT, defined as participants received ONO-7475 with a minimum dose intensity of 75% within DLT evaluation period [from first dose to Day 28] and had completed Day 28 assessments.
Measure: Count of Participants; unit: Participants
Groups:
- ONO-7475 Total (Part A): Part A ONO-7475 evaluable data, total
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg | ONO-7475 Total (Part A)
Number analyzed (Participants) | 10 | 3 | 7 | 20
Participants
  Numbers of participants experienced DLT | 0 | 0 | 0 | 0
  Numbers of participants not experienced DLT | 10 | 3 | 7 | 20

9. Secondary Outcome: Pharmacokinetics (Cmax and Ctrough) of ONO-7475 (Part A)
Description: Part A Pharmacokinetics Cmax of ONO-7475 assessed on day 1 and day 28, and Ctrough of ONO-7475 assessed on day 28 (pre-dose).
Time Frame: Day 1 and Day 28
Population: Pharmacokinetic (PK) analysis set, in participants who received at least 1 dose of ONO-7475 and with evaluable PK parameter resulted were summarised.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg
Number analyzed (Participants) | 7 | 3 | 6
ng/mL
  Cmax (ng/mL) day 1: number analyzed (Participants) | 7 | 1 | 6
  Cmax (ng/mL) day 1 | 90.8 (17.49) | 86 | 319.8 (73.99)
  Cmax (ng/mL) day 28: number analyzed (Participants) | 1 | 2 | 2
  Cmax (ng/mL) day 28 | 369.0 | 189.5 (96.87) | 1037 (229.58)
  Ctrough (ng/mL) day 28: number analyzed (Participants) | 4 | 3 | 5
  Ctrough (ng/mL) day 28 | 192.7 (154.23) | 353.0 (347.89) | 588.4 (250.90)

10. Secondary Outcome: Pharmacokinetics (Tmax) of ONO-7475 (Part A)
Description: Part A Pharmacokinetics Tmax of ONO-7475 assessed on day 1 and day 28.
Time Frame: Day 1 and Day 28
Population: Pharmacokinetic (PK) analysis set, in participants who received at least 1 dose of ONO-7475 and with evaluable PK parameter resulted were summarised. Insufficient evaluable data available for day 28 Tmax values in 3 mg dose group.
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg
Number analyzed (Participants) | 7 | 2 | 6
Hour (h)
  Tmax (h) day 1: number analyzed (Participants) | 7 | 1 | 6
  Tmax (h) day 1 | 3.5 (2.18) | 5.6 | 3.2 (2.4)
  Tmax (h) day 28: number analyzed (Participants) | 0 | 2 | 3
  Tmax (h) day 28 |  | 1.5 (2.12) | 4.3 (3.22)

11. Secondary Outcome: Pharmacokinetics (AUC) of ONO-7475 (Part A)
Description: Part A Pharmacokinetics (AUC0-10h) of ONO-7475 assessed on day 1 and day 28, (AUC0-24h) of ONO-7475 assessed on day 1.
Time Frame: Day 1 and Day 28
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg
Number analyzed (Participants) | 9 | 3 | 7
ng*h/mL
  AUC(0-10h) (ng*h/mL) day 1 | 559.3 (247.66) | 649.3 (296.73) | 2086.2 (767.91)
  AUC(0-10h) (ng*h/mL) day 28: number analyzed (Participants) | 1 | 2 | 3
  AUC(0-10h) (ng*h/mL) day 28 | 2534 | 1124.9 (654.75) | 6202.5 (2406.09)
  AUC(0-24h) (ng*h/mL) day 1: number analyzed (Participants) | 7 | 1 | 6
  AUC(0-24h) (ng*h/mL) day 1 | 1358.4 (198.56) | 1506.9 | 4870.3 (1147.48)

12. Secondary Outcome: Pharmacokinetics (T1/2) of ONO-7475 (Part A)
Description: Part A Pharmacokinetics T1/2 of ONO-7475 assessed on day 1 and day 28. T1/2 was not calculable due to insufficient evaluable data.
Time Frame: Day 1 and Day 28
Population: Pharmacokinetic (PK) analysis set, in participants who received at least 1 dose of ONO-7475 and with evaluable PK parameter resulted were summarised. T1/2 was not calculable due to insufficient evaluable data.
Groups:
- ONO-7475 3 mg: Part A initial dose level
- ONO-7475 6 mg: Part A 2nd dose level
Arm/Group | ONO-7475 3 mg | ONO-7475 6 mg | ONO-7475 10mg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Pharmacokinetics of the Food Effect on ONO-7475 (Part A)
Description: Part A Pharmacokinetics (Cmax, Tmax, AUC, T1/2, Ctrough) of the food effect on ONO-7475 assessed as ratio of Day57/Day28 and comparing pharmacokinetic parameters from dosing under fasted and non-fasted conditions assessed in 6mg and 10mg dose groups.
Time Frame: Day 28 and Day 57
Population: Pharmacokinetic analysis set, in participants who received at least 1 dose of ONO-7475 and with evaluable PK parameter results. Food effect was not evaluated in 3mg dose group. Tmax, T1/2 and Ctrough ratios were not calculable due to insufficient data.
Measure: Median (Full Range); unit: ratio
Arm/Group | ONO-7475 3 mg | ONO-7475 6mg | ONO-7475 10mg
Number analyzed (Participants) | 0 | 1 | 1
ratio
  Day 57/Day 28 ratio of Cmax |  | 0.89 [0.89 to 0.89] | 1.13 [1.13 to 1.13]
  Day 57/Day 28 ratio of AUC (0-10h) |  | 0.88 [0.88 to 0.88] | 1.69 [1.69 to 1.69]

14. Secondary Outcome: Pharmacodynamics (Axl and Mer Inhibition) of ONO-7475 (Part A)
Description: Assessment of the pharmacodynamic activity by measurement of Axl and Mer inhibition using a Plasma Inhibitory Activity (PIA) assay. PIA is a flow cytometry assay measuring auto-phosphorylation in Axl-expressing Ba/F3 and Mer-expressing Ba/F3 cells, respectively the percentage of inhibition. Pre-dose samples were collected for the analysis on day 2 and day 28.
Time Frame: Day 2 and Day 28
Population: Pharmacodynamic (PD) analysis set, in participants who received at least 1 dose of ONO-7475 and with evaluable PD parameter results were summarised.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10mg
Number analyzed (Participants) | 6 | 1 | 5
percentage
  Axl %inhibition Day 2 Pre-dose: number analyzed (Participants) | 6 | 1 | 3
  Axl %inhibition Day 2 Pre-dose | 53.13 (20.971) | 19.10 (NA) — SD not calculable | 88.57 (4.876)
  Axl %Inhibition Day 28 Pre-Dose: number analyzed (Participants) | 3 | 1 | 2
  Axl %Inhibition Day 28 Pre-Dose | 82.50 (11.811) | 99.5 (NA) — SD not calculable | 90.30 (8.344)
  Mer %inhibition Day 2 Pre-dose: number analyzed (Participants) | 2 | 0 | 5
  Mer %inhibition Day 2 Pre-dose | 31.40 (9.475) |  | 55.78 (11.932)
  Mer %Inhibition Day 28 Pre-Dose: number analyzed (Participants) | 1 | 1 | 3
  Mer %Inhibition Day 28 Pre-Dose | 42.60 (NA) — SD not calculable | 69.1 (NA) — SD not calculable | 91.5 (10.209)

15. Secondary Outcome: Overall Response Rate and Duration of Response in ONO-7475 Groups (Part A)
Description: Part A analysis of best overall response. Duration of response analysis was not performed as no response of complete remission, Morphologic complete remission with incomplete blood count recovery, morphologic leukemia-free state, or partial remission was observed.
Time Frame: From baseline up to maximum of 32 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10 mg | Total
Number analyzed (Participants) | 10 | 3 | 7 | 20
Participants
  Complete response | 0 | 0 | 0 | 0
  Morphologic complete remission with incomplete blood count recovery | 0 | 0 | 0 | 0
  Morphologic leukemia-free state | 0 | 0 | 0 | 0
  Partial remission | 0 | 0 | 0 | 0
  Treatment failure | 5 | 3 | 5 | 13
  Not evaluated / assessed | 5 | 0 | 2 | 7

16. Secondary Outcome: Event Free Survival in ONO-7475 Groups (Part A)
Description: Part A analysis of event free survival in ONO-7475 treatment groups
Time Frame: From baseline up to maximum of 32 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ONO-7475 3mg | ONO-7475 6mg | ONO-7475 10 mg | Total
Number analyzed (Participants) | 10 | 3 | 7 | 20
Months | 1.0 [0.3 to 1.3] | 0.9 [0.9 to 1.6] | 0.9 [0.9 to 1.6] | 1.0 [0.9 to 1.1]

17. Secondary Outcome: Pharmacokinetics (Cmax) of ONO-7475 in Treatment Group ONO-7475 + Venetoclax (Part D)
Description: Part D Pharmacokinetics (Cmax) of ONO-7475 in treatment group ONO-7475 + venetoclax.
Time Frame: Day 29
Population: Pharmacokinetic (PK) analysis set, in participants who received at least 1 dose of ONO-7475 and with evaluable PK parameter results.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ONO-7475 6mg + Venetoclax: Part D combination treatment group of ONO-7475 6mg + venetoclax
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 15
ng/mL | 622 (236)

18. Secondary Outcome: Pharmacokinetics (Tmax) of ONO-7475 in Treatment Group ONO-7475 + Venetoclax (Part D)
Description: Part D Pharmacokinetics (Tmax) of ONO-7475 in treatment group ONO-7475 + venetoclax.
Time Frame: Day 29
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 15
Hour (h) | 5.58 (5.84)

19. Secondary Outcome: Pharmacokinetics (AUC) of ONO-7475 in Treatment Group ONO-7475 + Venetoclax (Part D)
Description: Part D Pharmacokinetics (AUC) of ONO-7475 in treatment group ONO-7475 + venetoclax.
Time Frame: Day 29
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 15
ng*h/mL
  AUC (0-10h) (ng*h/mL) of ONO-7475 Day 29 | 4810 (1990)
  AUC (0-24h) (ng*h/mL) of ONO-7475 Day 29 | 11100 (4820)

20. Secondary Outcome: Pharmacokinetics (T1/2) of ONO-7475 in Treatment Group ONO-7475 + Venetoclax (Part D)
Description: Part D Pharmacokinetics (T1/2) of ONO-7475 in treatment group ONO-7475 + venetoclax.
Time Frame: Day 29
Population: Pharmacokinetic (PK) analysis set, in participants who received at least 1 dose of ONO-7475 and with evaluable PK parameter results. T1/2 of ONO-7475 was not calculable due to insufficient evaluable data.
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 0

21. Secondary Outcome: Pharmacokinetics (Cmax) of Venetoclax in Treatment Group ONO-7475 + Venetoclax (Part D)
Description: Part D Pharmacokinetics (Cmax) of Venetoclax in treatment group ONO-7475 + Venetoclax.
Time Frame: Day 1 and Day 29
Population: Pharmacokinetic (PK) analysis set, in participants who received at least 1 dose of venetoclax and with evaluable PK parameter results.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 17
ng/mL
  Cmax (ng/mL) Day 1 | 310 (281)
  Cmax (ng/mL) Day 29: number analyzed (Participants) | 15
  Cmax (ng/mL) Day 29 | 1870 (846)

22. Secondary Outcome: Pharmacokinetics (Tmax) of Venetoclax in Treatment Group ONO-7475 + Venetoclax (Part D)
Description: Part D Pharmacokinetics (Tmax) of Venetoclax in treatment group ONO-7475 + venetoclax.
Time Frame: Day 1 and Day 29
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 22
Hour (h)
  Tmax day 1: number analyzed (Participants) | 17
  Tmax day 1 | 6.72 (1.99)
  Tmax day 29: number analyzed (Participants) | 15
  Tmax day 29 | 7.07 (4.85)

23. Secondary Outcome: Pharmacokinetics (AUC) of Venetoclax in Treatment Group ONO-7475 + Venetoclax
Description: Part D Pharmacokinetics (AUC) of Venetoclax in treatment group ONO-7475 + venetoclax.
Time Frame: Day 1 and Day 29
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 22
ng*h/mL
  AUC (0-10h) day 1: number analyzed (Participants) | 17
  AUC (0-10h) day 1 | 1330 (1220)
  AUC (0-10h) day 29: number analyzed (Participants) | 15
  AUC (0-10h) day 29 | 14700 (8650)
  AUC (0-24h) day day 29: number analyzed (Participants) | 15
  AUC (0-24h) day day 29 | 32900 (19200)

24. Secondary Outcome: Pharmacokinetics (T1/2) of Venetoclax in Treatment Group ONO-7475 + Venetoclax (Part D)
Description: Part D Pharmacokinetics (T1/2) of Venetoclax in treatment group ONO-7475 + venetoclax.
Time Frame: Day 29
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 1
Hour (h) | 5.8

25. Secondary Outcome: Incidence of Adverse Events in ONO-7475 + Venetoclax Group (Part D)
Description: Part D Incidence (frequency > 20%) and severity (CTCAE grades) of treatment-emergent adverse events in ONO-7475 + Venetoclax Group, in preferred terms coded MedDRA version 23.1.
  CTCAE = common terminology criteria for adverse events (CTCAE) version 4.03.
Time Frame: as for outcome 5
Population: Safety analysis set, in participants who received at least 1 dose of ONO-7475 and/or venetoclax.
Measure: Count of Participants; unit: Participants
Groups:
- ONO-7475 6 mg + Venetoclax (All Grade); ONO-7475 6 mg + Venetoclax (Grade >/=3): Part D treatment group of ONO-7475 6 mg + Venetoclax
Arm/Group | ONO-7475 6 mg + Venetoclax (All Grade) | ONO-7475 6 mg + Venetoclax (Grade >/=3)
Number analyzed (Participants) | 22 | 22
Participants
  Participants with treatment-emergent adverse events | 21 | 20
  Fatigue | 10 | 0
  Diarrhoea | 7 | 0
  Febrile neutropenia | 7 | 7
  Hypophosphataemia | 7 | 0
  Anaemia | 6 | 5
  Nausea | 6 | 0
  Constipation | 5 | 0
  Headache | 5 | 0
  Hypokalaemia | 5 | 0
  Thrombocytopenia | 5 | 5
  Vomiting | 5 | 0

26. Secondary Outcome: Incidence of Serious Adverse Events in ONO-7475 + Venetoclax Group (Part D)
Description: Part D Incidence (frequency ≥ 2 participants) and severity (CTCAE grades) of serious treatment-emergent adverse events in ONO-7475 + Venetoclax Group (Part D), preferred term coded with MedDRA version 23.1.
  CTCAE = Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: as for outcome 5
Population: Safety analysis set, in participants who received at least 1 dose of ONO-7475 and/or venetoclax
Measure: Count of Participants; unit: Participants
Groups:
- ONO-7475 6mg + Venetoclax (All Grades); ONO-7475 6mg + Venetoclax (≥ Grade 3): Part D ONO-7475 6mg + Venetoclax
Arm/Group | ONO-7475 6mg + Venetoclax (All Grades) | ONO-7475 6mg + Venetoclax (≥ Grade 3)
Number analyzed (Participants) | 22 | 22
Participants
  Participants with serious adverse events | 13 | 13
  Sepsis | 3 | 3
  Febrile neutropenia | 7 | 7
  Gastrointestinal hemorrhage | 2 | 2

27. Secondary Outcome: Overall Response Rate in ONO-7475 + Venetoclax Group (Part D)
Description: Part D Summary of best overall response in ONO-7475 + Venetoclax group.
Time Frame: From baseline up to maximum of 21 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Groups:
- ONO-7475 6mg + Venetoclax (Part D): Part D ONO-7475 6mg + venetoclax group
Arm/Group | ONO-7475 6mg + Venetoclax (Part D)
Number analyzed (Participants) | 22
Participants
  Complete remission | 0
  Complete remission with incomplete hematologic recovery | 1
  Morphologic leukemia free state | 1
  Partial remission | 2
  Treatment failure | 16
  Not evaluated / assessed | 2

28. Secondary Outcome: Duration of Response in ONO-7475 + Venetoclax Group (Part D)
Description: Part D Duration of response in ONO-7475 6mg + Venetoclax group.
Time Frame: From baseline up to maximum of 21 months
Population: Full analysis set. Participants with best response assessed as complete remission, complete remission with partial hematologic recovery, complete remission with incomplete hematologic recovery, morphologic leukemia free state and partial remission were included in analysis.
Measure: Mean (Standard Deviation); unit: Months
Groups:
- ONO-7475 6mg + Venetoclax: Part D ONO-7475 6mg + Venetoclax
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 4
Months | 1.881 (2.5073)

29. Secondary Outcome: Event-Free Survival and Overall Survival in ONO-7475 + Venetoclax Group (Part D)
Description: Part D analysis of event free survival and overall survival in ONO-7475 6mg + Venetoclax group
Time Frame: From baseline up to maximum of 21 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 22
Months
  Event free survival | 0.99 [0.95 to 1.9]
  Overall survival | 4.01 [2.60 to 10.25]

30. Secondary Outcome: Transfusion Independence Rate (Part D)
Description: Part D analysis of transfusion Independence rate. Rate of maintenance of transfusion independence = percentage of patients who were transfusion independent post-baseline based upon the patients who were transfusion independent at baseline.
  Calculated using the Clopper-Pearson method.
Time Frame: From baseline up to maximum of 21 months
Population: Full analysis set and in participants who were transfusion independent at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ONO-7475 6mg + Venetoclax
Number analyzed (Participants) | 7
percentage of participants | 87.5 [47.3 to 99.7]

ADVERSE EVENTS:
Time Frame: From an onset date on or after study drug start date and no later than 30 days after permanent discontinuation of study drug or initiation of new anti-cancer therapy, whichever occurs first (maximum 32 months for Part A and 21 months for Part D).
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Groups:
- ONO-7475 3mg (Part A): Part A ONO-7475 initial dose level 3mg
- ONO-7475 6mg (Part A): Part ONO-7475 2nd dose level 6mg
- ONO-7475 10mg (Part A): Part A ONO-7475 3rd dose level 10mg
- ONO-7475 6mg + Venetoclax (Part D): Part D combination of ONO-7475 6mg + venetoclax
Arm/Group | ONO-7475 3mg (Part A) | ONO-7475 6mg (Part A) | ONO-7475 10mg (Part A) | ONO-7475 6mg + Venetoclax (Part D)
All-Cause Mortality (participants affected / at risk) | 10/10 | 3/3 | 5/7 | 15/22
Serious Adverse Events (participants affected / at risk) | 9/10 | 2/3 | 6/7 | 13/22
Other Adverse Events (participants affected / at risk) | 10/10 | 3/3 | 7/7 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-7475 3mg (Part A) (N=10) | ONO-7475 6mg (Part A) (N=3) | ONO-7475 10mg (Part A) (N=7) | ONO-7475 6mg + Venetoclax (Part D) (N=22)
Pneumonia (Infections and infestations) | 3 | 1 | 0 | 0
Sepsis (Infections and infestations) | 3 | 1 | 0 | 3
Klebsiella bacteraemia (Infections and infestations) | 2 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Stenotrophomonas sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex oesophagitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 4 | 7
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-7475 3mg (Part A) (N=10) | ONO-7475 6mg (Part A) (N=3) | ONO-7475 10mg (Part A) (N=7) | ONO-7475 6mg + Venetoclax (Part D) (N=22)
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 2 | 7
Vomiting (Gastrointestinal disorders) | 5 | 2 | 2 | 5
Nausea (Gastrointestinal disorders) | 3 | 2 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 5
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral mucosa haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Poor dental condition (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Post-tussive vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 3 | 2 | 2 | 10
Oedema peripheral (General disorders) | 4 | 2 | 1 | 3
Pyrexia (General disorders) | 2 | 0 | 2 | 3
Asthenia (General disorders) | 0 | 1 | 1 | 2
Chills (General disorders) | 0 | 1 | 1 | 0
Generalised oedema (General disorders) | 1 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 5
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 3
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0
Muscle abscess (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Stenotrophomonas sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Systemic candida (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 2 | 5
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 4
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 2
White blood cell count increased (Investigations) | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
Blood lactic acid increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 4
Retinogram abnormal (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 3 | 2 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cataract cortical (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0
Night blindness (Eye disorders) | 1 | 0 | 0 | 2
Retinal aneurysm (Eye disorders) | 0 | 1 | 0 | 0
Retinal thickening (Eye disorders) | 1 | 0 | 0 | 0
Retinopathy (Eye disorders) | 1 | 0 | 0 | 0
Scleral haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 3
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2 | 3
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Leukaemic retinopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial prior to submission for publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT03176277/Prot_SAP_000.pdf